CLINICAL TRIAL: NCT01893164
Title: Comparison of Simple Decompression Versus Anterior Subcutaneous and Intramuscular Transposition of the Ulnar Nerve for Moderate and Severe Cubital Tunnel Syndrome ：A Randomized Double-blind Control Trial
Brief Title: Comparison of Different Surgical Treatments for Different Scales of Cubital Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Rui Li, chief doctor and PhD supervisor, Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JilinU-218-RLi
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Cubital Tunnel Syndrome
Keywords: cubital tunnel syndrome; simple decompression; anterior subcutaneous transposition of ulnar nerve; anterior intramuscular transposition of ulnar nerve; severity scale
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- moderate cubital tunnel syndrome (Experimental): Sensory,Intermittent paresthesias; vibratory perception normal or decreasedMotor,Measurable weakness in pinch or grip strengthTests,Elbow flexion test or Tinel's sign is positive; finger crossing may be abnormal.Treated by simple decompression,anterior subcutaneous transposition and anterior intramuscular transposition of the ulnar nerve.
  Interventions: Procedure: simple decompression; Procedure: anterior subcutaneous transposition; Procedure: anterior intramuscular transposition
- severe cubital tunnel syndrome (Experimental): Sensory,Persistent paresthesias; vibratory perception decreased; abnormal two-point discrimination(static >6 mm, moving >4 mm)Motor,Measurable weakness in pinch and grip plus muscle atrophyTests,Positive elbow flexion test or positive Tinel's sign may be present; finger crossing usually abnormal.Treated by simple decompression,anterior subcutaneous transposition and anterior intramuscular transposition of the ulnar nerve.
  Interventions: Procedure: simple decompression; Procedure: anterior subcutaneous transposition; Procedure: anterior intramuscular transposition

INTERVENTIONS:
Procedure: simple decompression — decompression of the ulnar nerve
  Other Names: SDP
Procedure: anterior subcutaneous transposition — transposition of the ulnar nerve into subcutaneous bed
  Other Names: ASCT
Procedure: anterior intramuscular transposition — transposition of the ulnar nerve into muscular tissue
  Other Names: AIMT

SUMMARY:
The purpose of this study is to determine which is the best surgery to treat different severity scales of cubital tunnel syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to determine which one of the simple decompression,anterior subcutaneous and intramuscular transposition of the ulnar nerve has the best outcomes for moderate and severe cubital tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed cubital tunnel syndrome
* moderate and severe cubital tunnel syndrome.

Exclusion Criteria:

* Significant cervical spine and shoulder disease
* deformity or distortion of the cubital tunnel due to previous trauma to elbow
* recurrent cubital tunnel syndrome after previous surgery
* mild cubital tunnel syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
sensation | at 6 months post-operatively
  Sensory disturbance were tested with Semmes-Weinstein filaments and sensory deficits were categorized according to the Yale sensory scale. According to standard scoring system that designed, the severity of sensation and function of the ulnar nerve was scored as follows: ---- 0, Abscent sensation; 1, Decrease or abnormal sensation; 2, Intact sensation.

SECONDARY OUTCOMES:
Muscle strength | at 6 months post-operatively
  Muscle strength was evaluated with the grading system from the Medical Research Council which is based upon a scale of zero to five: 0, No muscle contraction; 1,Flicker or trace of muscle contraction; 2,Limb or joint movement possible only with gravity eliminated; 3,Limb or joint movement against gravity only; 4,Power decreased but limb or joint movement possible against resistance; 5,Normal power against resistance. Then results were scored as follows: ---- 0,Poor (0-1); 1,Moderate (2-3); 2,Good (4-5)
pain | at 6 months post-operatively
  Visual Analogue Scale (VAS) with scores of zero to ten (0 for no pain and 10 intolerable pain) then scored as follows: ---- 0, Sever (8-10); 1, Slight (4-7); 2, none (0-3)
electromyography | at 6 months post-operatively
  Compare the result at 6 months post-operatively with the result before operation.To see if there is an improvement in the function of the ulnar nerve.0,no improvement;1,improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, chief doctor, Study Chair — Hand Sugery Department of the China-Japan Union Hospital
Locations (1):
- Hand Surgery Department of China-Japan Union Hospital, Changchun, Jilin, China